CLINICAL TRIAL: NCT03154580
Title: Marijuana Cue-Reactivity & Seeking Behavior in Regular Cannabis Users: A Pilot Test of Glutamatergic Modulation
Brief Title: Marijuana Cue-Reactivity & Seeking Behavior in Regular Cannabis Users
Acronym: MCN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Leslie Lundahl, Principal Investigator, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MCN-1
Record Dates: First submitted 2017-04-25; First posted 2017-05-16 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Marijuana Abuse
MeSH Terms: conditions — Marijuana Abuse | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- N-acetylcysteine 0mg X Cue Exposure (neutral) (Placebo Comparator)
  Interventions: Drug: N-acetyl cysteine
- N-acetylcysteine 0mg X Cue Exposure (marijuana) (Placebo Comparator)
  Interventions: Drug: N-acetyl cysteine
- N-acetylcysteine 2400mg X Cue Exposure (neutral) (Active Comparator)
  Interventions: Drug: N-acetyl cysteine
- N-acetylcysteine 2400mg X Cue Exposure (marijuana) (Active Comparator)
  Interventions: Drug: N-acetyl cysteine

INTERVENTIONS:
Drug: N-acetyl cysteine — Participants will receive 4 capsules at 11:15am on each experimental session day.

SUMMARY:
The purpose of the proposed study is to examine the relationship between marijuana reminders, or "cues", craving for marijuana, and marijuana use. The principal investigator is also assessing whether N-acetylcysteine, can reduce marijuana craving or use.

DETAILED DESCRIPTION:
This study involves three screening sessions that could last about 3 hours each.

Part of this study will be conducted on an inpatient unit where the participant will live for 4 straight nights.

During the inpatient stay participants will participant in experimental sessions where they will be asked to smoke cigarettes containing either marijuana or placebo (a blank). Participants will be asked to take capsules that could contain N-acetylcysteine or placebo (blank).

Participants will be asked to complete questionnaires and have vital signs (blood pressure, heart rate) monitored.

Participants will be asked to participate in overnight sleep recordings, a polysomnogram (PSG).

ELIGIBILITY:
Inclusion Criteria:

* Participants will be healthy individuals 21-55 year olds who use marijuana.
* Marijuana use will be verified by self-report and THC-positive urine samples. -Participants must meet DSM 5 criteria for Cannabis Use Disorder and be willing to participate in research but not seeking treatment.

Exclusion Criteria:

* Candidates with the following conditions will be excluded:
* Serious psychiatric illness (e.g. psychotic or bipolar disorder
* Recent (past 5 years) suicide attempts
* Major depression that is not substance-induced)
* Substance Use Disorders (SUD) other than Cannabis or Nicotine Use Disorders and Mild Alcohol Use Disorder
* Neurological diseases (e.g. stroke, seizures)
* Cardiovascular problems (e.g. myocardial infarction, angina, systolic BP >160 or <95 mmHg, diastolic BP >95 mmHg, clinically abnormal ECG)
* Pulmonary diseases (e.g. asthma, TB)
* Systemic diseases (e.g. hepatitis, autoimmune, Cushing syndrome)
* Cognitive impairment (<80 IQ)
* Past-month exposure to medications that increase study risk (e.g. toxicity to major organs, asthma inhalers)
* Women who are pregnant (urine HCG), lactating (self-report), or if heterosexually active and not using (self-report) medically approved birth control measures (oral/depot contraceptives, IUD, condom/foam, sterilization, tubal ligation)
* Seeking treatment for a Substance Use Disorder.
* Individuals unable to give voluntary informed consent will be excluded. Applicants interested in treatment will be excluded from the study and referred to a treatment program.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Marijuana Craving Visual Analog Scale (VAS) (Self-report measure) | Change is being assessed. Marijuana Craving VAS administered at baseline 0900, at 0930, 1000, 1030, 1100, 1230, 1250, 1310, 1320, 1330, 1345, 1400, 1430, 1500, 1530, and 1600.
Marijuana Craving Questionnaire (Self-report measure) | Change is being assessed. Marijuana Craving Quest.administered at baseline 0900, at 0930, 1000, 1030, 1100, 1230, 1345, 1400, 1430, 1500, 1530, and 1600.
Marijuana Rating Form (Self-report measure) | Change is being assessed. Marijuana Rating Form administered at baseline 0900, at 0930, 1000, 1030, 1100, 1230, 1345, 1400, 1430, 1500, 1530, and 1600.
Subjective Effects Scale Visual Analog Scale (VAS) (Self-report measure) | Change is being assessed. Subjective Effects Scale administered at baseline 0900, at 0930, 1000, 1030, 1100, 1230, 1345, 1400, 1430, 1500, 1530, and 1600.
Questionnaire of Smoking Urges (Self-report measure) | Change is being assessed. Questionnaire is administered at baseline 0900, at 0930, 1000, 1030, 1100, 1230, 1345, 1400, 1430, 1500, 1530, and 1600.
Marijuana Withdrawal Checklist | Change is being assessed. Questionnaire is administered at baseline 0900, at 0930, 1000, 1030, 1100, 1230, 1345, 1400, 1430, 1500, 1530, and 1600.
NAC Side Effect Checklist | Change is being assessed. Questionnaire is administered at baseline 0900, at 0930, 1000, 1030, 1100, 1230, 1345, 1400, 1430, 1500, 1530, and 1600.
Systolic blood pressure (physiological effects) | Change is being assessed. Systolic blood pressure measured at baseline 0900, at 0930, 1000, 1030, 1100, 1230, 1345, 1400, 1430, 1500, 1530, and 1600.
Diastolic blood pressure (physiological effects) | Change is being assessed. Diastolic blood pressure measured at baseline 0900, at 0930, 1000, 1030, 1100, 1230, 1345, 1400, 1430, 1500, 1530, and 1600.
Heart rate (physiological effects) | Change is being assessed. Heart rate measured at baseline 0900, at 0930, 1000, 1030, 1100, 1230, 1345, 1400, 1430, 1500, 1530, and 1600.
Core-body temperature (physiological effects) | Change is being assessed. Core-body temperature measured at baseline 0900, at 0930, 1000, 1030, 1100, 1230, 1345, 1400, 1430, 1500, 1530, and 1600.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Lundahl, PhD, Principal Investigator — Wane State University
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No